CLINICAL TRIAL: NCT07175168
Title: Prevalence of Translocation Phenotyping in Children With Down Syndrome and Their Parents: A Cross-Sectional Study
Brief Title: Prevalence of Translocation Phenotyping in Children With Down Syndrome and Their Parents
Acronym: PTP-DS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Bassem, resident, Assiut University
Other Study IDs: DS-TRANSLOC-2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Translocation Down Syndrome; Chromosomal Abnormalities
Keywords: Balanced translocation; trisomy 21; Translocation; Down syndrome
MeSH Terms: conditions — Chromosome Aberrations; Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — "Peripheral blood samples will be collected from children and their parents for cytogenetic (karyotype) analysis. Samples will be processed for standard cytogenetic testing and retained only as required for completion/verification of the cytogenetic analyses. No specimens will be used for future unspecified DNA research or biobanking unless additional ethics approval is obtained and separate written consent is obtained from the participant/parent."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Down Syndrome: Children (0-18 years) with cytogenetically confirmed Down syndrome, recruited from Assiut University Children's Hospital and Health Insurance Hospital. All participants will undergo full clinical assessment and karyotyping.
  Interventions: Other: No medical or experimental intervention will be administered
- Parents of Children with Down Syndrome: Available biological parents of enrolled children will undergo chromosomal analysis (karyotyping) to determine balanced translocation carrier status.
  Interventions: Other: No medical or experimental intervention will be administered

INTERVENTIONS:
Other: No medical or experimental intervention will be administered — Laboratory procedures (blood sampling for karyotyping, basic investigations such as echocardiography, thyroid function tests, abdominal ultrasound) are part of standard diagnostic assessment, not rese

SUMMARY:
This research study will investigate a special type of Down syndrome called translocation Down syndrome. While most children with Down syndrome have an extra copy of chromosome 21, about 3-4% have this extra chromosome material attached to another chromosome, known as a translocation. This form can sometimes be inherited from a parent who carries a balanced translocation.

The aim of the study is to find out how common translocation Down syndrome is among children with confirmed Down syndrome in Assiut, Egypt, and to check whether their parents are carriers of a balanced translocation. Understanding this will help improve family counseling, estimate the chance of recurrence in future pregnancies, and guide genetic screening and prevention strategies.

DETAILED DESCRIPTION:
Down syndrome (DS) is the most common chromosomal disorder, occurring in approximately 1 in 700 live births worldwide, and is associated with intellectual disability and multiple congenital anomalies. The majority of cases (about 95%) are due to free trisomy 21, while translocation DS accounts for 3-4% and mosaic DS for 1-2%. Translocation DS occurs when extra chromosome 21 material is attached to another chromosome, commonly chromosome 14 or 22. This form is clinically important because it may be inherited from a balanced translocation carrier parent, which has major implications for recurrence risk, genetic counseling, and family planning.

This cross-sectional descriptive study will be conducted at Assiut University Children's Hospital, Pediatric Genetics Unit, and Health Insurance Hospital from October 2025 to September 2027. A total of 230 children with cytogenetically confirmed Down syndrome will be included, along with their available parents for karyotyping. Children with free trisomy 21 or mosaicism will be excluded.

Data collection will include demographic characteristics, detailed family and medical history, full clinical examination, and cytogenetic analysis of both children and their parents. Baseline investigations such as echocardiography, thyroid function tests, and abdominal ultrasound will be performed to document associated comorbidities.

The primary outcome is the prevalence of unbalanced translocation among children with Down syndrome. The secondary outcome is the prevalence of balanced translocation carrier status among parents. Data analysis will be performed using SPSS v27 with descriptive and inferential statistics, with significance set at p < 0.05.

Ethical approval has been obtained from the Assiut University Faculty of Medicine Ethics Committee. Written informed consent will be secured from all parents prior to participation.

This study is expected to provide valuable local prevalence data on translocation Down syndrome, support genetic counseling efforts, and inform recommendations for parental karyotyping and recurrence risk assessment in Egyptian families affected by Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years with confirmed diagnosis of Down syndrome by chromosomal analysis.

Availability of at least one biological parent willing to undergo chromosomal analysis.

Exclusion Criteria:

* Children with Down syndrome due to free trisomy 21 or mosaicism.

Incomplete parental data or refusal of parental participation.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cytogenetically confirmed Down syndrome attending Assiut University Children's Hospital and Health Insurance Hospital, along with their biological parents for karyotyping.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of unbalanced translocation Down syndrome among children with cytogenetically confirmed Down syndrome | At the time of enrollment (October 2025 - September 2027)
  Proportion of enrolled children (0-18 years) with unbalanced translocation identified by standard karyotyping.

IPD SHARING:
Plan to Share IPD: Undecided